CLINICAL TRIAL: NCT05053880
Title: A Phase 1b/2a Study of ACT001 and Anti-PD-1 in Patients With Surgically Accessible Recurrent Glioblastoma Multiforme
Brief Title: A Study to Evaluate Safety and Efficacy of ACT001 and Anti-PD-1 in Patients With Surgically Accessible Recurrent Glioblastoma Multiforme
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Accendatech USA Inc. (Industry)
Collaborators: C3 Research Associates (Unknown); Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACT001-US-001
Record Dates: First submitted 2021-08-12; First posted 2021-09-23 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Recurrent Glioblastoma Multiforme(GBM)
Keywords: GBM; Brain; Blastoma; Neoplasm
MeSH Terms: conditions — Glioblastoma; Neoplasms | interventions — ACT001; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Phase 1b dose exploration will enroll up to a maximum of 18 patients. Phase 2a, randomized/2-treatment arm part, will enroll up to 30 patients in two treatment arms. Arm A (treatment with Pembrolizumab) will enroll 10 patients. Arm B (treatment with the combination ACT001 plus Pembrolizumab) will enroll 20 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1b dose exploration (Experimental): 1b dose exploration for 18 patients - The starting dose of ACT001 will be administered in combination with a single intravenous (IV) infusion of Pembrolizumab. After recovery from surgical resection, dosing will resume on a 3 weekly cycle and will consist of Pembrolizumab (standard dosing) and daily ACT001. Evaluation of a dose level of at least three (3) patients after completing one cycle of treatment post-surgery is required prior to commencing the next dose level.
  Interventions: Drug: ACT001
- 2a- Randomized/Two-treatment Arm (Experimental): 30 Patients will be randomized to Arm A or Arm B at a ratio of 1 (Arm A) : 2 (Arm B). 10 patients will be randomized to the Pembrolizumab only arm (Arm A) and 20 patients will be randomized to the ACT001 plus Pembrolizumab arm (Arm B).
  Interventions: Drug: ACT001 + Pembrolizumab

INTERVENTIONS:
Drug: ACT001 — Phase1b - Starting approximately 2 weeks prior to the scheduled surgery, patient will receive an assigned dose of ACT001 by mouth in combination with a single dose of 200 mg pembrolizumab via an intravenous (IV-through a tube in vain) infusion in the clinic. Then patient will self administer ACT001 capsules twice daily by mouth, at the dose to which patient is assigned, until the evening prior to scheduled surgery. Patient will then undergo surgery to remove all or part of tumor. This a standard 3+3 dose escalation.
  Arms: 1b dose exploration
Drug: ACT001 + Pembrolizumab — Phase 2a - Starting approximately 2 weeks prior to the scheduled surgery, patient will receive a single dose of 200 mg pembrolizumab via an intravenous (IV) infusion in the clinic (an IV infusion means the drug will be delivered through a tube in your vein). Patient will then self-administer ACT001 capsules twice daily by mouth, at the dose to which patient is assigned, until the evening prior to scheduled surgery. Patient then will undergo surgery to remove all or part of tumor.
  Arms: 2a- Randomized/Two-treatment Arm

SUMMARY:
The current design provides a window to analyze the impact of the ACT001+Pembrolizumab combination on the tumor microenvironment and disease outcomes.

DETAILED DESCRIPTION:
Phase 1b: The identified RP2D of combined ACT001 with Pembrolizumab will be determined by standard 3+3 dose escalation methodology among three ACT001 dosages (200mg, 400mg and 800mg, BID) with standard Pembrolizumab dosage. Patients will be dosed approximately 2 weeks prior to surgical resection with a single dose of Pembrolizumab and ACT001. Tumor resection will be performed and a biopsy will be obtained from the resected tumor tissue to evaluate the impact of the study drugs on the TME. After recovery from surgery, patients will resume ACT001 and Pembrolizumab until tumor progression (assessed by iRANO) or an AE requiring discontinuation of study drug. The Safety Monitoring Committee (SMC) will review the data available from all evaluable patients at each dose level prior to recommending escalation to the next dose level.

Phase 2a: Using the same dosing schedule and ACT001 dosage as determined in Phase 1b. Patients will be randomized to receive either Pembrolizumab only treatment (Arm A, 10 patients) or ACT001 plus Pembrolizumab treatment (Arm B, 20 patients).

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided written informed consent.
2. ≥ 18 years old at time of screening visit.
3. Histologically confirmed GBM at the time of diagnosis.
4. First or second relapse by the time of consenting.
5. Tumor progression (magnetic resonance imaging [MRI], defined by RANO) post prior treatments.
6. Feasibility for re-surgery.
7. Karnofsky Performance Status ≥ 70% (requires occasional assistance, but able to care for most of their needs, equivalent to < ECOG 2).
8. Must be ≥ 4 weeks from administration of last dose of cancer therapy (including radiation therapy or chemotherapy). The patient must have recovered from all treatment-related toxicities to less than grade 2 per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
9. Life expectancy of ≥ 3 months.
10. Adequate organ function (absolute neutrophil count ≥1.5 x 109 /L, lymphocytes ≥ 0.5 x 109 /L, platelets ≥ 75 x 109 /L, hemoglobin ≥ 10 g/dl; total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤ 5.0 x ULN if liver metastasis); plasma creatinine ≤ 1.5 x ULN; QTc < 450 ms (male), < 470 ms (female).
11. Female patients are eligible if they are of:

    1. Non-childbearing potential, defined as

       * Previous hysterectomy or bilateral oophorectomy
       * Previous bilateral tubal ligation
       * Post-menopausal (total cessation of menses for ≥ 1 year)
    2. Childbearing potential with a negative serum pregnancy test at screening (within 7 days of the first investigational product administration) and uses a highly effective method contraception before study entry and throughout the study until 28 days after the last investigational product administration. Highly effective contraception (<1% failure rate per year), when used consistently and in accordance with both the product label and the instructions of the physician, are defined as follows:

       * Vasectomized partner who is sterile prior to the female patient's enrolment and is her sole sexual partner
       * An intrauterine device with a documented failure rate of less than 1% per year
       * Double barrier contraception defined as condom with a female diaphragm
12. Male patients, if sexually active, must agree to use a highly effective method of contraception (< 1% failure rate per year) with their female partners from screening until 28 days following the last study drug administration.
13. Absence of deteriorating neurological symptoms, new onset of seizures and the need for increasing doses of corticosteroids.
14. Absence of toxicity from prior therapy (excluding alopecia) that has not resolved to ≤ Grade 1 unless otherwise specified.
15. Absence of other clinically significant concomitant active medical disorder, based on the investigator's judgement

Exclusion Criteria:

1. The patient has uncontrolled infection.
2. The patient has serious diseases such as unstable angina pectoris, myocardial infarction in the past 6 months, heart failure (New York Heart Association class > II) or stroke within 6 months prior to the enrollment.
3. A gastrointestinal absorption disorder that would limit the bioavailability of oral drugs or if patient cannot take oral drugs.
4. Uncontrolled brain metastases or spinal cord compression. Patients who were treated with surgical resection or radiation therapy completing at least 4 weeks earlier are eligible if they are neurologically stable, not taking glucocorticoids and have a follow-up. MRI scan performed within the previous 4 weeks showing no tumor progression.
5. Pre-existing allergy to ACT001 or related compounds.
6. A patient has active autoimmune disease managed by systemic treatments in the past 2 years (i.e. the use of corticosteroids, immunosuppressive drugs or other disease modifying agents). Of note, a replacement therapy, e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, is not considered a form of systemic treatment.
7. A known history of, or any evidence of an active non-infectious pneumonitis.
8. Treatment with cancer therapies such as chemotherapy or radiation therapy either currently or within 4 weeks of ACT001 dosing. An exception is focal radiation for symptomatic bone metastases, which must not be within 2 weeks of ACT001 dosing.
9. History of treatment with immune CPB and Avastin (or other antiangiogenic or anti-vascular endothelial growth factor agents).
10. High dose of corticosteroids (> 4mg/day of dexamethasone or equivalent for at least 3 consecutive days) within two weeks of enrolment for GBM treatment.
11. A patient has received other systemic immunosuppressive treatments such as mTOR inhibitor everolimus four weeks prior to registration.
12. A patient has a diagnosis of ongoing immunodeficiency due to other diseases such as human immunodeficiency virus (HIV) infection.
13. Unresolved toxicity from prior antitumor therapy, defined as toxicities (excluding alopecia) that have not resolved to < Grade 2 as scored using the CTCAE current version. Exceptions may be allowed for stable toxicities after discussion with the investigator and sponsor.
14. Major surgery within 30 days of commencing first study therapy.
15. Pregnant or breast-feeding females.
16. A history of infection with HIV or hepatitis B or C viruses.
17. The patient has participated in other drug clinical studies < 4 weeks prior to obtaining the informed consent.
18. The patient is, in the opinion of the investigator, unsuitable for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
1b-Incidence, type and severity of treatment-emergent AEs (TEAEs) | Approximately 7 months. Each cycle is 21 days; from start of first dose with investigational product until completion of the last study related procedure (including follow-up for safety assessments- 30days after last dose)
1b-Dose limiting toxicities (DLTs) | From first dose of study therapy until the end of the first post-surgery cycle (Cycle 1, Day 21).
  A DLT is defined as any of the following
  * Haematological toxicity
    * Grade 4 neutropenia
    * Grade ≥ 3 febrile neutropenia or neutropenic infection
    * Grade 4 thrombocytopenia
    * Grade 3 thrombocytopenia with clinically significant bleeding
  * Non-haematological toxicity
    * Grade ≥ 3 nausea, vomiting or diarrhoea despite optimal supportive therapy
    * Grade ≥ 3 hypertension despite appropriate intervention
    * Other grade ≥ 3 non-haematological toxicity, except grade 3 fatigue or transient events (such as allergic reactions or electrolyte disturbances) that are readily controlled with medical therapy and/or are of no clinical concern
1b-Mean changes in vital sign measurements-Heart Rate | Approximately 8months/ patient. Each cycle is 21 days. Start at screening, Pre-surgical Treatment Period, Cycle 1 and each subsequent Cycle and 30 days after last dose
  Mean change from baseline in vital sign measurements reported in beats/min (inclusive) at each study timepoint.
1b-Mean changes in vital sign measurements- supine blood pressure | Approximately 8months/ patient.Each cycle is 21 days. Start at screening, Pre-surgical Treatment Period, Cycle 1 and each subsequent Cycle and 30 days after last dose
  Mean change from baseline in vital sign measurements reported in mmHg at each study timepoint
1b-Mean changes in vital sign measurements- body temperature | Approximately 8months/ patient. Each cycle is 21 days. Start at screening, Pre-surgical Treatment Period, Cycle 1 and each subsequent Cycle and 30 days after last dose
  Mean change from baseline in vital sign measurements reported in degrees Celsius (0C) at each study timepoint.
1b-Mean changes in vital sign measurements- respiratory rate | Approximately 8months/ patient. Each cycle is 21 days. Start at screening, Pre-surgical Treatment Period, Cycle 1 and each subsequent Cycle and 30 days after last dose
  Mean change from baseline in vital sign measurements reported in bpm at each study timepoint
1b-Mean changes in electrocardiogram (ECG) parameters | approximately 8months/patient. Each cycle is 21 days. Start at screening, Pre-surgical Treatment Period, Cycle 1 and each subsequent Cycle and 30 days after last dose
  Mean change from baseline in electrocardiogram (ECG) parameters of heart rate, ventricular rate, PR interval, QRS duration, and QTcF.
1b-Mean changes in Karnofsky Performance Scale score | Approximately 8 months/patient. Each cycle is 21 days. Start at screening, Pre-surgical Treatment Period, Cycle 1 and each subsequent Cycle and 30 days after last dose
  Mean change from baseline in Karnofsky Performance Scale score
2a-Progression free survival (PFS) at 6 months | Six months after initiation of study therapy

SECONDARY OUTCOMES:
1b-Incidence of DLTs according to the MTD/RP2D evaluation process. | From first dose of study therapy (per surgery) until the end of the first post-surgery cycle (Cycle 1, Day 21). Each cycle is 21 days.
1b- Pharmacokinetics (PK) of ACT001 in Plasma concentrations in tumor. | PK analysis will be collected on Day 1 of the pre surgical treatment period.
  Determine ACT001 trough levels in tumor samples.
2a-Overall survival | Approximately 7months/patient- screening period is not included. Cycle 1 Day 1 until death, loss to follow-up, withdrawal of consent, date of disease progression or whichever occurs first
  Overall survival (OS) is defined as time from start of ACT001 dosing at day 1 of cycle 1 until the date of death or date from any cause, assessed up to disease progression.
2a-Incidence, type and severity of TEAEs | From start of dosing until 30 days after the last dose of ACT001
  Summary of the treatment-emergent Adverse events experienced during treatment. Adverse events are assessed with Common Terminology Criteria for Adverse Events (CTCAE) 5.0. TEAEs are defined as any medical occurrence reported or observed after the start of dosing with investigational product until completion of the last study related procedure (including follow-up for safety assessments)
2a-Concentration of ACT001 in resected tumor biopsy tissue. | Tissue at Surgical Resection only.

CONTACTS AND LOCATIONS:
Overall Officials: Doug Cai, MD, Study Director — Accendatech USA Inc.
Locations (1):
- UT MD Anderson Cancer Center, Dept of Neuro-Oncology, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No